CLINICAL TRIAL: NCT05729464
Title: Risk Factors and Prediction Model of Cancer-associated Venous Thromboembolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yongsheng Jiang (Other)
Responsible Party: Sponsor-Investigator, Yongsheng Jiang, Department of Oncology ,Tongji Hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20221313
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Venous Thromboses; Neoplasms
MeSH Terms: conditions — Venous Thrombosis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer patients with venous thrombosis
- cancer patients without venous thrombosis

SUMMARY:
The purpose of this study is to identify risk factors of cancer-associated venous thrombosis and develop a prediction model to assist clinicians in tailoring anticoagulant therapy.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a prevalent complication in cancer patients. Compared with the general population, patients with tumors are four to seven times more likely to develop venous thrombotic events. A population-based cohort study showed that the incidence of VTE in these patients has increased steadily over the past decade. Cancer-associated thrombosis may result in discontinuation of antineoplastic therapy, decreased quality of life, and increased mortality. Clinical trials indicate that prophylactic anticoagulation leads to a significantly lower rate of thrombotic disorders. However, due to the fact that thromboprophylaxis treatment increases the risk of bleeding complications and that the risk of VTE varies widely among individuals, only patients at high risk of thrombosis will benefit from primary thromboprophylaxis. In this setting, the use of anticoagulant drugs is challenging. So, the purpose of this study is to identify risk factors of cancer-associated venous thrombosis and develop a prediction model to assist clinicians in tailoring anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* with a histological diagnosis of cancer.

Exclusion Criteria:

* received long-term anticoagulant therapy;
* without a clear primary site of malignancy;
* had a follow-up of fewer than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with malignant tumors in Tongji Hospital in Wuhan.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
cancer-associated venous thrombosis | 12 months since receiving anti-cancer therapy
  including deep venous thrombosis and pulmonary embolism

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: Undecided
If needed, we will share the study protocol, informed consent form and clinical study report.

REFERENCES:
- [Background] Mulder FI, Bosch FTM, van Es N. Primary Thromboprophylaxis in Ambulatory Cancer Patients: Where Do We Stand? Cancers (Basel). 2020 Feb 5;12(2):367. doi: 10.3390/cancers12020367. PMID 32033438
- [Background] Lloyd AJ, Dewilde S, Noble S, Reimer E, Lee AYY. What Impact Does Venous Thromboembolism and Bleeding Have on Cancer Patients' Quality of Life? Value Health. 2018 Apr;21(4):449-455. doi: 10.1016/j.jval.2017.09.015. Epub 2017 Nov 10. PMID 29680102
- [Background] Mahajan A, Brunson A, White R, Wun T. The Epidemiology of Cancer-Associated Venous Thromboembolism: An Update. Semin Thromb Hemost. 2019 Jun;45(4):321-325. doi: 10.1055/s-0039-1688494. Epub 2019 Apr 30. PMID 31041801
- [Background] Mulder FI, Horvath-Puho E, van Es N, van Laarhoven HWM, Pedersen L, Moik F, Ay C, Buller HR, Sorensen HT. Venous thromboembolism in cancer patients: a population-based cohort study. Blood. 2021 Apr 8;137(14):1959-1969. doi: 10.1182/blood.2020007338. PMID 33171494
- [Background] Fernandes CJ, Morinaga LTK, Alves JL Jr, Castro MA, Calderaro D, Jardim CVP, Souza R. Cancer-associated thrombosis: the when, how and why. Eur Respir Rev. 2019 Mar 27;28(151):180119. doi: 10.1183/16000617.0119-2018. Print 2019 Mar 31. PMID 30918022
- [Background] Riondino S, Ferroni P, Zanzotto FM, Roselli M, Guadagni F. Predicting VTE in Cancer Patients: Candidate Biomarkers and Risk Assessment Models. Cancers (Basel). 2019 Jan 15;11(1):95. doi: 10.3390/cancers11010095. PMID 30650562
- [Background] Kim AS, Khorana AA, McCrae KR. Mechanisms and biomarkers of cancer-associated thrombosis. Transl Res. 2020 Nov;225:33-53. doi: 10.1016/j.trsl.2020.06.012. Epub 2020 Jul 6. PMID 32645431
- [Background] Hisada Y, Mackman N. Cancer-associated pathways and biomarkers of venous thrombosis. Blood. 2017 Sep 28;130(13):1499-1506. doi: 10.1182/blood-2017-03-743211. Epub 2017 Aug 14. PMID 28807983
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292
- [Background] Key NS, Khorana AA, Kuderer NM, Bohlke K, Lee AYY, Arcelus JI, Wong SL, Balaban EP, Flowers CR, Francis CW, Gates LE, Kakkar AK, Levine MN, Liebman HA, Tempero MA, Lyman GH, Falanga A. Venous Thromboembolism Prophylaxis and Treatment in Patients With Cancer: ASCO Clinical Practice Guideline Update. J Clin Oncol. 2020 Feb 10;38(5):496-520. doi: 10.1200/JCO.19.01461. Epub 2019 Aug 5. PMID 31381464
- [Background] Mulder FI, Candeloro M, Kamphuisen PW, Di Nisio M, Bossuyt PM, Guman N, Smit K, Buller HR, van Es N; CAT-prediction collaborators. The Khorana score for prediction of venous thromboembolism in cancer patients: a systematic review and meta-analysis. Haematologica. 2019 Jun;104(6):1277-1287. doi: 10.3324/haematol.2018.209114. Epub 2019 Jan 3. PMID 30606788